CLINICAL TRIAL: NCT07109128
Title: The T1D Talks Pilot Study: An Online Teen / Tween Group About Life With T1D and Managing the Emotions That Come With it
Brief Title: The T1D Talks Pilot Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Western Michigan University School of Medicine (Other)
Collaborators: Nemours Children's Health System (Other)
Responsible Party: Principal Investigator, Rachel Wasserman, Associate Professor, Western Michigan University School of Medicine
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: WMED1378; 11-23-JDFBMH-03 (Other Grant/Funding Number: American Diabetes Association)
Record Dates: First submitted 2025-04-23; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: adolescents; emotion regulation; group; virtual
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Emotional Regulation | interventions — Polysorbates

STUDY DESIGN:
Intervention Model Description: 3 sequential trials of a novel behavioral intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The T1D Talks Virtual Group Intervention for Teens and Tweens with T1D (Experimental): Experimental: The T1D Talks Group Intervention. This is the intervention, as this is a proof of concept pilot study, we will only have an intervention arm.
  Interventions: Behavioral: The T1D Talks: A Virtual Group for Teens and Tweens with T1D

INTERVENTIONS:
Behavioral: The T1D Talks: A Virtual Group for Teens and Tweens with T1D — The T1D Talks intervention is an 11 session, virtual (online), group intervention. The T1D Talks intervention teaches developmentally appropriate emotion regulation (ER) skills and facilitates practicing these skills via role-plays and in-session experiences that are meant to elicit strong emotions. The investigators adapted the content and situations of an established intervention to be relevant for youth with T1D (e.g., practicing ER skills while role playing situations like telling parents about high blood glucose numbers or telling a coach about needing to take a time out from a game because of a low blood glucose level). The intervention also provides basic diabetes education about risky situations (e.g., how physical activity can affect blood glucose).

SUMMARY:
Despite recent technological advances in type 1 diabetes (T1D) treatment, adolescents are the only age group for which glycemic levels have not improved. Technology and education help adolescents execute the mechanics of managing blood glucose levels, but do not help adolescents manage the emotional distress that arises when T1D management goals conflict with social/emotional goals (e.g., taking insulin for a meal in front of new friends vs. trying to "fit-in"). The emotional distress caused by such situations can be difficult to manage and can lead to unhealthy risk behaviors and disengagement in T1D self-management (e.g., deciding to skip a lunch-time bolus to avoid bolusing in front of new friends).

A novel approach in T1D research is to target emotions directly by promoting emotion regulation skills. In the general population, emotion regulation interventions have demonstrated success in preventing both unhealthy behaviors and mood disorders among younger adolescents, including younger adolescents with social-emotional risk-factors like low SES. The investigators' scientific premise is that an emotion regulation intervention for younger adolescents with T1D (age 12-14) could promote skills to help youth manage emotional burdens of living with T1D, reduce unhealthy and risky T1D self-management behaviors, and prevent unhealthy patterns of behaviors and distress/mood disorders that often appear in later adolescence.

Using the ORBIT Model, a systematic framework for developing behavioral interventions for people with chronic diseases, the investigators adapted an evidence-based, manualized emotion regulation intervention for young adolescents, so that it is relevant for youth with T1D. The current study is a natural extension of this previous work. For the current study, the investigators propose to complete a feasibility and acceptability trial of this novel emotion regulation intervention for youth with T1D.

The investigators aimed to pilot the novel emotion regulation intervention (11 virtual group sessions) with 3 sequential groups of 6-8 young adolescents (age 12-14) with T1D in each group and obtain feedback from facilitators and participants and their parents after each session, and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* T1D for at least 1 year
* the ability to read/write and converse in English
* reliable internet connection and a virtual meeting capable device (tablet or laptop)

Exclusion Criteria:

* a chronic medical condition that requires intensive daily management
* a significant mental health or cognitive disability that would prevent them from participating

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-11-14 (Estimated); Study Completion 2025-11-14 (Estimated)

PRIMARY OUTCOMES:
Percent of participants who attended the intervention | Through study completion, up to 12 weeks
  Feasibility will be demonstrated by average individual participation in at least 70% of the sessions, and >70% of participants completing the intervention by participating in the last session.
Percent of participants who rated each session as acceptable | Through study completion, up to 12 weeks
  The percentage of participants who rated each session as "acceptable" on a post-session survey rating scales that were developed for this study. 6 items on the session evaluation survey assess the following: relevance, trust in the information, ease of understanding, learning novel information, and interest in topics. Item responses include a 5-point Likert scale from "strongly disagree to strongly agree". The research team will average participant's responses across the items, thus total score could be a minimum of 1 and a maximum of 5, with a higher score indicating higher acceptability of the intervention. The intervention will be considered acceptable if ≥ 70% of participants rate each session as acceptable, as indicated by a total score >3.
Percent of participants who rated the overall intervention as acceptable | Through study completion, up to 12 weeks
  The percentage of participants who rated the intervention, as a whole, as "acceptable" on a post-intervention survey rating scales that were developed for this study. 16 items on the intervention evaluation survey assess, one's perceptions of the intervention. Item responses include a 5-point Likert scale from "strongly disagree to strongly agree". The research team will reverse score items that negatively worded and average participant's responses across the items, thus total score could be a minimum of 1 and a maximum of 5, with a higher score indicating higher acceptability of the intervention. The intervention will be considered acceptable if ≥ 70% of participants rate the intervention as acceptable, as indicated by a total score >3.

SECONDARY OUTCOMES:
Difficulties in Emotion Regulation- Short Form Scale | Baseline to post-intervention, up to 11 weeks
  The change in the DERS-SF will be measured from baseline to post-intervention (up to 11 weeks). Self-report measure of emotion regulation strategies of particularly negative emotions, rated on a 5 point scale, with higher score indicating greater engagement in strategies.
Emotion Regulation Behaviors Scale (ERBS-R) | Baseline to post-intervention, up to 11 weeks
  The change in the ERBS-R will be measured from baseline to post-intervention (up to 11 weeks). The ERBS-R measures the use of the specific emotion regulation strategies taught in the ER intervention. Using a scale of 1 ("never") to 5 ("all of the time"), with higher scores indicate more frequent use of the strategies taught.
Implicit Theories of Emotion Scale- Child Version (ITES-C) | Baseline to post-intervention, up to 11 weeks
  The change in the ITES-C will be measured from baseline to post-intervention (up to 11 weeks). The ITES-C Self subscale assessed adolescents' beliefs about the controllability of their emotions. Six items were rated on a 6-point scale from "strongly disagree" to "strongly agree" and were averaged to create a score. Higher scores indicate stronger beliefs in an incremental theory of emotion (that emotions are malleable) as opposed to an entity theory (that emotions are fixed).
Affect Dysregulation Scale (ADS) | Baseline to post-intervention, up to 11 weeks
  The change in the ADS will be measured from baseline to post-intervention (up to 11 weeks). The ADS assesses the frequency of adolescents' difficulties with affect regulation, with a higher score indicating greater difficulty.
Early Adolescent Temperament Questionnaire (EATQ-R select subscales) | Baseline to post-intervention, up to 11 weeks
  The change in the EATQ-R will be measured from baseline to post-intervention (up to 11 weeks), including the following subscales: 5 subscales (29 items): Activation Control , Attention, Frustration , Inhibitory Control, and Surgency. The ADS assesses the frequency of adolescents' difficulties with affect regulation, with a higher score indicating greater difficulty. The current questionnaire has been designed to specifically tap experiences common to adolescents, and is available in self- and parent-report formats. It assesses temperament and self-regulation via adaptation of scales used in studies of children and adults.
Problem Areas in Diabetes: Teen (PAID-T) | Baseline to post-intervention, up to 11 weeks
  The change in the PAID-T will be measured from baseline to post-intervention (up to 11 weeks). The PAID-T is a 26-item self-report measure of diabetes-specific emotional distress in teens with diabetes, rated on a 6 point scale, with higher scores indicating greater distress.
Diabetes-related Executive Functioning Scale- short form (DREFS-SF) | Baseline to post-intervention, up to 11 weeks
  The change in the DREFS-SF will be measured from baseline to post-intervention (up to 11 weeks). The DREFS-SF is an 11-item self-report and parent proxy screening measure to assess behaviors related to diabetes- specific executive functioning, with higher scores indicating greater difficulty.
Diabetes-Specific Risk-Taking Inventory (DSRI) | Baseline to post-intervention, up to 11 weeks
  The change in the DSRI will be measured from baseline to post-intervention (up to 11 weeks). The DSRI is a 31-item (+3 items for insulin pump users) self-report measure assessing risky T1D self-management behaviors, rated on a 6 point scale, with higher score indicating more frequent engagement in risky diabetes-related health behaviors.
Diabetes Knowledge Questionnaire (DKQ) | Baseline to post-intervention, up to 11 weeks
  The change in the DKQ will be measured from baseline to post-intervention (up to 11 weeks). The DKQ is adapted from other, established diabetes knowledge questionnaires for the purpose of this study. Higher scores indicate more accurate knowledge of information related to diabetes management.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Wasserman, PhD, Principal Investigator — Western Michigan University Homer Stryker MD School Of Medicine
Locations (1):
- Nemours Children's Hospital, Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified and cleaned, item-level spreadsheet data for all variables will be shared with other researchers (along with example quantifications and transformations from initial raw data) via deposit in the data sharing repositories. The rationale for sharing only cleaned data is to foster ease of data reuse. Aggregate survey datasets and summaries of debriefing sessions, containing no identifiers, data collection instruments, codebook and data dictionary, qualitative analysis protocols, and code and statistical analysis protocols will be freely available via the data sharing repository (below).
Time Frame: The investigators will share this data by May 2027, either within 6 months of publication or within 18 months of the conclusion of the funding period (November 14, 2025), if the study remains unpublished.
Access Criteria: Public use and restricted access study data and associated documentation will be made available to the research community free of charge through openICPSR, (https://www.openicpsr.org/openicpsr/) which is a self-publishing repository for social, behavioral, and health sciences research data.